CLINICAL TRIAL: NCT01959165
Title: MEDI7183 Phase 2 Study in Japanese Ulcerative Colitis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5172C00001
Record Dates: First submitted 2013-10-08; First posted 2013-10-09 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-04

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis, Japanese, subcutaneously
MeSH Terms: conditions — Colitis, Ulcerative | interventions — abrilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- MEDI7183 dose 1 (Experimental): Double blinded
  Interventions: Drug: MEDI7183 low dose
- MEDI7183 dose 2 (Experimental): Double blinded
  Interventions: Drug: MEDI7183 medium dose
- MEDI7183 dose 3 (Experimental): Double blinded
  Interventions: Drug: MEDI7183 high dose
- Placebo (Placebo Comparator): Double blinded
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: MEDI7183 low dose — MEDI7183 will be administered by SC on Day 1, Week 2, 4, and 8
  Arms: MEDI7183 dose 1
Drug: MEDI7183 medium dose — MEDI7183 will be administered by SC on Day 1, Week 2, 4, and 8
  Arms: MEDI7183 dose 2
Drug: MEDI7183 high dose — MEDI7183 will be administered by SC on Day 1, and placebo for MEDI7183 at Week 2, 4, and 8
  Arms: MEDI7183 dose 3
Drug: Matching Placebo — Placebo will be administered by SC on Day 1, Week 2,4, and 8
  Arms: Placebo

SUMMARY:
This is a multi-centre, randomised, double-blind, placebo controlled, parallel group, Phase II study to evaluate efficacy and safety of 3 doses of MEDI7183, in Japanese subjects with moderate to severe UC

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Diagnosis of UC established by clinical and endoscopic evidence and corroborated by a histopathology report
* Moderate to severe active UC as defined by a total Mayo score of 6 to 12 with rectosigmoidoscopy score ≥ 2 during screening period
* Demonstrated an inadequate response to, loss of response to, or intolerance to at least one of immunomodulators or Anti- TNF-α agents. etc.

Exclusion Criteria:

* Disease limited to the rectum
* Toxic megacolon
* Crohn's Disease
* History of subtotal colectomy with ileorectostomy or colectomy with ileoanal pouch, Koch pouch, or ileostomy for UC
* Planned bowel surgery within 12 weeks from Visit 2
* Stool positive for C. difficile toxin at screening
* Primary Sclerosing Cholangitis
* History of gastrointestinal surgery within 8 weeks of Visit 2
* Any uncontrolled or clinically significant systemic disease
* Condition or disease that, in the opinion of the investigator would pose a risk to subject safety or interfere with study evaluation, procedures or completion
* Subjects with positive HBsAg, HBsAb, HBcAb or HCVAb serology at screening etc

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-11-21 (Actual); Primary Completion 2015-08-11 (Actual); Study Completion 2018-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toshifumi Hibi, Director and Professor, Principal Investigator — Centre for Advanced IBD Research and Treatment, Kitasato Institute Hospital, Kitasato University; Ki Rito, Study Physician, Study Director — AztraZeneca, Tokyo, Japan
Locations (20):
- Japan (20):
  - Research Site, Chikushino-shi
  - Research Site, Fujiidera-shi
  - Research Site, Fukuyama-shi
  - Research Site, Hamamatsu
  - Research Site, Kagoshima
  - Research Site, Kamakura-shi
  - Research Site, Kyoto
  - Research Site, Minatoku
  - Research Site, Morioka
  - Research Site, Niigata
  - Research Site, Nishinomiya-shi
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Sakura-shi
  - Research Site, Sapporo
  - Research Site, Sayama-shi
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
  - Research Site, Yokkaichi-shi
  - Research Site, Yokohama

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the protocol part, the number of enrolled participants was 44. This number means 44 participants who were assigned and received the treatment. In fact, 59 participants signed informed consent form. Out of the enrolled, 45 participants were assigned, and 1 out of the 45 participants discontinued the study without receiving any treatment.
Pre-assignment Details: Out of the 59 enrolled participants, 14 participapatients were not assigned to any arm. Out of these 14 participants, 13 participants did not meet the eligibility criteria and 1 participants withdrew the informed consent.
Groups:
- Placebo: placebo double blind phase
- MEDI7183 21 mg: MEDI7183 21 mg double blind phase
- MEDI7183 70 mg: MEDI7183 70 mg double blind phase
- MEDI7183 210 mg: MEDI7183 210 mg double blind phase
Period: Overall Study
Arm/Group | Placebo | MEDI7183 21 mg | MEDI7183 70 mg | MEDI7183 210 mg
Started | 13 | 11 (1 patient discontinued the study without any treatment out of 11 patients.) | 12 | 9
Completed (completed patients number in double blind period) | 12 | 10 | 12 | 7
Not Completed | 1 | 1 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — overdose | 0 | 0 | 0 | 1
Not completed — Welfare recipient | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: In MEDI7183 21 mg arm, 11 patients were randomised, but 1 patient discontinued the study without any treatment. Therefore, this patient was excluded from all of the analyses in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI7183 21 mg | MEDI7183 70 mg | MEDI7183 210 mg | Total
Number analyzed (Participants) | 13 | 10 | 12 | 9 | 44
Age, Continuous [Mean (Full Range); unit: Years] | 38.0 [20 to 64] | 45.9 [22 to 63] | 39.8 [19 to 62] | 33.1 [22 to 57] | 39.3 [19 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 4 | 3 | 15
  Male | 8 | 7 | 8 | 6 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 13 | 10 | 12 | 9 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
duration of Ulcerative Colitis [Mean (Full Range); unit: years] | 5.41 [1.0 to 8.5] | 6.75 [0.8 to 21.8] | 5.43 [1.3 to 11.8] | 3.29 [0.6 to 7.8] | 5.28 [0.6 to 21.8]
use of 5-aminosalicylates [Count of Participants; unit: Participants] — use of 5-aminosalicylates at baseline of double-blind phase
  Participants
    Number of participants who took the drug | 11 | 10 | 10 | 8 | 39
use of oral corticosteroids [Count of Participants; unit: Participants] — use of oral corticosteroids at baseline of double blind phase
  Participants
    Number of paticipants who took the drug | 3 | 1 | 3 | 2 | 9
use of immunomodulators [Count of Participants; unit: Participants] — use of immunomodulators at baseline of double blind phase
  Participants
    Number of participants who took the drug | 7 | 3 | 8 | 5 | 23
any prior use of anti-TNF-a agents [Count of Participants; unit: Participants]
  Number of participants who took the drug | 8 | 5 | 7 | 6 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Remission at Week 8
Description: Remission at Week 8 was defined as a total Mayo score 2 points or smaller, and with no individual subscore more than 1 point.
Time Frame: 8 weeks
Population: All randomised participants who received at least one dose of investigational drug during the double-blind phase
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI7183 21 mg | MEDI7183 70 mg | MEDI7183 210 mg
Number analyzed (Participants) | 13 | 10 | 12 | 9
Participants
  Number of participants with Remission | 0 | 1 | 2 | 1

2. Secondary Outcome: Number of Participants With Response at Week 8
Description: Response at Week 8 was assessed by total Mayo score. Response was defined as decrease 3 points or more and 30 percents in total Mayo score compared to baseline, and with an accompanying decrease in the subscore for rectal bleeding of 1 point or more, or with an absolute subscore for rectal bleeding of 0 or 1.
Time Frame: 8 weeks
Population: All randomised participants who received at least one dose of investigational drug during the double-blind phase
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI7183 21 mg | MEDI7183 70 mg | MEDI7183 210 mg
Number analyzed (Participants) | 13 | 10 | 12 | 9
Participants
  Number of participants with Response | 7 | 3 | 6 | 6

3. Secondary Outcome: Number of Participants With Mucosal Healing at Week 8
Description: Mucosal healing was defined as an absolute Mayo subscore for rectosigmoidoscopy of 0 or 1.
Time Frame: 8 weeks
Population: All randomised participants who received at least one dose of investigational drug during the double-blind phase
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI7183 21 mg | MEDI7183 70 mg | MEDI7183 210 mg
Number analyzed (Participants) | 13 | 10 | 12 | 9
Participants
  Number of participants with Mucosal healing | 4 | 1 | 4 | 4

4. Secondary Outcome: Number of Participants With Response at Week 12
Description: Response at Week 12 was assessed by Partial Mayo Score. Response was defined as reduction by 2 or more points and 25% in Partial Mayo Score compared to baseline.
Time Frame: 12 weeks
Population: All randomised participants who received at least one dose of investigational drug during the double-blind phase
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI7183 21 mg | MEDI7183 70 mg | MEDI7183 210 mg
Number analyzed (Participants) | 13 | 10 | 12 | 9
Participants
  Number of participants with Response | 6 | 3 | 6 | 6

ADVERSE EVENTS:
Time Frame: 12 weeks for DB period.
Description: AEs were collected after dosing. SAEs were collected after consent date.
Groups:
- Placebo: placebo double blind period
- MEDI7183 70 mg: MEDI7183 70 mg double blind period
- MEDI7183 210 mg: MEDI7183 210 mg double blind period
Arm/Group | Placebo | MEDI7183 21 mg | MEDI7183 70 mg | MEDI7183 210 mg
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/10 | 0/12 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/10 | 0/12 | 1/9
Other Adverse Events (participants affected / at risk) | 9/13 | 6/10 | 6/12 | 3/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | MEDI7183 21 mg (N=10) | MEDI7183 70 mg (N=12) | MEDI7183 210 mg (N=9)
colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — No other AEs were observed in the subject suffered this SAE.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | MEDI7183 21 mg (N=10) | MEDI7183 70 mg (N=12) | MEDI7183 210 mg (N=9)
nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 3 (3) | 2 (2)
colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
enterocolitis viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
injection site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
white blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
skin swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less